CLINICAL TRIAL: NCT04510844
Title: A Phase IV, Double-Blind, Placebo-Controlled, Multi-Center Trial To Study The Effects Of Evolocumab In Stage IV-V Chronic Kidney Disease: The Cardiovascular and Lipid-Lowering Effects Of Evolocumab In Advanced Chronic Kidney Disease Trial
Brief Title: Evolocumab In Advanced Chronic Kidney Disease Trial
Acronym: EVO-CKD
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: loss of funding
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-00405; 21-00455 (Other: NYU Langone Health)
Record Dates: First submitted 2020-06-30; First posted 2020-08-12 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Chronic Kidney Diseases; High Cholesterol
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypercholesterolemia | interventions — evolocumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Study Drug Group (Experimental): Participants who will receive a shot of the Evolocumab at Visit 3 and self-administer the rest of the shots at visit 4-7.
  Interventions: Drug: Evolocumab
- Placebo group (Placebo Comparator): Participants who will receive a Placebo shot at Visit 3 and self-administer the rest of the shots at visit 4-7.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Evolocumab — Evolocumab is commercially available in the United States and is manufactured by Amgen. Drug and placebo, will be supplied by the manufacturer. The SureClick® pre-filled auto injector contain Evolocumab (140 mg) acetate (1.2 mg), polysorbate 80 (0.1 mg), proline (25 mg) in water for Injection. Evolocumab will be administered at a dose of 420 mg subcutaneously once monthly.
  Arms: Study Drug Group
Other: Placebo — Placebo will be supplied by the manufacturer. Placebo auto injectors will be identically packaged but will lack the active ingredient. Placebo will be administered at an equivalent volume to Evolocumab and given subcutaneously once monthly.
  Arms: Placebo group

SUMMARY:
110 individuals with stage 4-5 Chronic Kidney Disease (CKD) will be randomized to 1-year of blinded Evolocumab or placebo. Subjects will undergo evaluation of circulating lipids at baseline and end of study. A substudy including 50 subjects will assess myocardial rest and stress positron emission tomography (PET) at baseline and at 1-year.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of evolocumab (Repatha®)-a Food and Drug Administration (FDA)-approved biological drug that has been shown to reduce LDL cholesterol (bad cholesterol) Early data show that the beneftis of evolocumab may be increased as kidney function declines. This trial is therefore designed to provide additional evidence regarding the safety and cholesterol-lowering effects of evolocumab compared with placebo, a pill that has no therapeutic effect, in advanced CKD patients.

ELIGIBILITY:
Inclusion Criteria:

* CKD Stage 4-5 defined as

  * eGFR ≤30 mL/min/1.73m2 on screening lab OR
  * Treatment with maintenance hemodialysis for at least 30 days prior to screening
* LDL ≥70 mg/dL and

  * Treatment with maximal tolerated doses of a statin OR
  * Statin intolerance defined as any history of intolerance or allergy to ≥1 statin
* Age 40-80 years

  * Individuals ≤60 years old are required to have ≥1 of the following cardiovascular risk factors:

    * History of CV disease
    * History of peripheral vascular disease
    * Diabetes
    * Smoking
    * Baseline LDL ≥160 mg/dL
    * Macroalbuminuria (albumin to creatinine ratio ≥300 mg/g on spot sample)

Exclusion Criteria:

* Age >80 years
* Expected survival < 1 year
* Transplant expected within < 1 year
* Active liver disease (history of cirrhosis, ALT or AST > 2x ULN)
* CPK > 5x ULN at screening
* Malignancy within 5 years except for non-melanoma skin cancers, cervical in-situ carcinoma, breast ductal carcinoma in situ, or stage 1 prostate carcinoma
* Subject has received drugs that are strong inhibitors of cytochrome P-450 3A4 within 1 month prior to randomization or is likely to require such treatment during the study period
* Currently enrolled in another interventional study
* Female subject who has not used at least (1) effective method of birth control for at least 1 month prior to screening or (2) is not willing to use such a method during treatment and for an additional 15 weeks after the end of treatment, unless the subject is sterilized or postmenopausal.

  * Effective measures of birth control include surgical sterilization, barrier methods, hormonal contraceptives and intrauterine devices.
* Pregnant or breast-feeding subjects
* Known sensitivity or intolerance to study medications

The following additional criteria will be utilized to exclude individuals from participating in the PET substudy:

* Severe asthma or obstructive lung disease defined by

  * Hospitalization for asthma or obstructive lung disease within 8 weeks
  * Use of oral steroids for lung disease within 8 weeks
  * Chronic oxygen therapy
  * Use of rescue inhalers ≥three times weekly in the previous 4 weeks
* History of seizures
* Second or third-degree AV block, unless a functioning pacemaker is present
* Sinus node dysfunction unless a functioning pacemaker is present

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Absolute change in LDL cholesterol concentration | Baseline, Week 52
  The primary endpoint is selected to evaluate the key pharmacologic mechanism underlying Evolocumab's cardiovascular benefits. This will be analyzed with Lipid parameters.

SECONDARY OUTCOMES:
Number of Serious Adverse Events (SAEs) | Baseline, Week 52
Change in coronary flow reserve (CFR) | Baseline, Week 52
  Change in coronary flow reserve (CFR), the key secondary efficacy endpoint, is a measure of overall cardiovascular health.This test provides an integrative measure of myocardial microvascular supply and myocardial endothelial function as well as large vessel coronary flow. Change in coronary flow reserve over one year as measured by cardiac PET scanning.

CONTACTS AND LOCATIONS:
Overall Officials: David Charytan, MD, Principal Investigator — NYULangone Health
Locations (2):
- United States (2):
  - NYU Langone Nephrology Associates - Long Island, Mineola, New York
  - NYU Langone Health, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data.Upon reasonable request. Requests should be directed to David.charytan@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.